CLINICAL TRIAL: NCT07086391
Title: A Prospective Clinical Study on Different Methods of Aerosolized Polymyxin B Inhalation for the Treatment of Carbapenem-Resistant Gram-Negative Bacterial Pneumonia
Brief Title: Different Methods of Aerosolized Polymyxin B Inhalation for Treating Carbapenem-Resistant Gram-Negative Bacterial Pneumonia.
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Lili Zhou, Associate Chief Physician, Fujian Medical University Union Hospital
Other Study IDs: 2022YF033-03
Record Dates: First submitted 2025-04-14; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-04

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; Pneumonia - Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 25mg polymyxin B + 5ml sterile water via jet nebulizer (respirator-assisted).
  Interventions: Device: Polymyxin B Sulfate 25mg Jet Nebulization / Vibrating Mesh Nebulization
- Group B: 25mg polymyxin B + 5ml sterile water via vibrating mesh nebulizer (respirator-assisted).
  Interventions: Device: Polymyxin B Sulfate 25mg Jet Nebulization / Vibrating Mesh Nebulization

INTERVENTIONS:
Device: Polymyxin B Sulfate 25mg Jet Nebulization / Vibrating Mesh Nebulization — * Group A: 25mg polymyxin B sulfate dissolved in 5ml sterile water, administered via jet nebulizer under mechanical ventilation.
  * Group B: 25mg polymyxin B sulfate dissolved in 5ml sterile water, administered via vibrating mesh nebulizer under mechanical ventilation.

SUMMARY:
Study Design:

A randomized, open-label, parallel-group clinical trial comparing the efficacy and safety of jet nebulization versus vibrating mesh nebulization of sulfate polymyxin B in mechanically ventilated patients with carbapenem-resistant Gram-negative bacterial pneumonia.

Participants:

144 patients (72 per group) will be enrolled from December 2023 to December 2025.

Interventions:

Group A: 25mg polymyxin B + 5ml sterile water via jet nebulizer (respirator-assisted).

Group B: 25mg polymyxin B + 5ml sterile water via vibrating mesh nebulizer (respirator-assisted).

Both groups receive additional intravenous polymyxin B (2.0mg/kg loading dose, followed by 1.25mg/kg every 12h) starting 12h after nebulization.

Treatment duration: 14 days.

Key Procedures:

Nebulization parameters: Fixed ventilator settings (SIMV+PSV mode, tidal volume 8ml/kg, PEEP 6cmH₂O).

Bronchoalveolar lavage (BAL) and blood sampling:

BAL fluid (BALF) and blood collected pre-nebulization (baseline), 1h post-nebulization, and at steady-state (days 3-7).

BALF analyzed for polymyxin B concentration, urea nitrogen, and inflammatory mediators (IL-6, TNF-α, etc.).

Primary Outcomes:

Clinical efficacy:

Total response rate (cure + improvement). 28-day survival rate. Time to fever resolution and bacterial clearance.

Drug exposure:

Polymyxin B concentration in alveolar epithelial lining fluid (ELF) and blood.

Secondary Outcomes:

Inflammatory response: Changes in BALF and serum IL-6, TNF-α, CRP levels.

Safety:

Nephrotoxicity (changes in serum creatinine/urea nitrogen). Airway complications (bronchospasm incidence).

Assessment Timeline:

Clinical monitoring: Daily evaluation of vital signs, sputum volume, and ventilator parameters.

Lab tests: Blood tests (hematology, renal function, inflammatory markers) at baseline, days 3/7/14.

Microbiological evaluation: Sputum cultures on days 3/7/14.

Statistical Analysis:

Efficacy and safety endpoints compared between groups using t-tests or chi-square tests.

A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia diagnosed per Chinese Thoracic Society criteria (radiographic + clinical evidence).
* Sputum culture-confirmed carbapenem-resistant Gram-negative bacteria susceptible to polymyxin B.
* ≥3 days of aerosolized polymyxin B therapy.
* Mechanically ventilated with an artificial airway.

Exclusion Criteria:

* Polymyxin B aerosol use planned for <3 days.
* Terminal status (life expectancy <48h).
* Severe liver/kidney dysfunction (ALT/AST >5× ULN; eGFR <30 mL/min).
* No informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated adults with carbapenem-resistant Gram-negative bacterial pneumonia (e.g., Pseudomonas aeruginosa) confirmed by sputum culture and susceptible to polymyxin B. Participants must receive ≥3 days of aerosolized polymyxin B via endotracheal tube/tracheostomy. Exclusions: life expectancy <48h, severe liver/kidney dysfunction, or lack of informed consent.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | Baseline (pre-treatment); End of Treatment (EOT, 14 days after starting polymyxin B)
  Percentage of patients with cure or improvement based on symptom resolution, microbiological clearance, and radiographic findings.

SECONDARY OUTCOMES:
28-Day Survival Rate | Baseline (pre-treatment); End of Treatment (EOT, 28 days after starting polymyxin B)
  Survival status assessed at 28 days post-treatment initiation.
Microbiological Clearance Rate | Baseline (pre-treatment); End of Treatment (EOT, 14 days after starting polymyxin B)
  Eradication or replacement of carbapenem-resistant pathogens.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No